CLINICAL TRIAL: NCT03223922
Title: Preservation of Cognition and Neuropsychiatric Functioning With Corpus Callosum Genu-Sparing Whole Brain Radiation Therapy for Brain Metastases: A Pilot Study
Brief Title: Neurocognitive Functioning With Genu-Sparing Whole Brain Radiation Therapy for Brain Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1737; IRB00128471 (Other: JHM IRB)
Record Dates: First submitted 2017-07-12; First posted 2017-07-21 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Brain Metastases
Keywords: whole brain radiation therapy; genu of corpus callosum; cognitive function
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be treated to a total dose of 30 Gy with a once daily fractionation schedule of 3 Gy per fraction, administered five days per week.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Corpus Callosum Genu-Sparing Whole Brain Radiation Therapy (Experimental): Genu-sparing whole brain radiation therapy (GS-WBRT) 30 Gy in 3 Gy per fraction
  Interventions: Radiation: whole brain radiation therapy

INTERVENTIONS:
Radiation: whole brain radiation therapy — Corpus Callosum Genu-Sparing Whole Brain Radiation Therapy Genu-sparing whole brain radiation therapy (GS-WBRT) 30 Gy in 3 Gy per fraction
  Other Names: WBRT

SUMMARY:
This is a trial that evaluates the preservation of cognition and neuropsychiatric function following genu-sparing whole brain radiation in patients with brain metastases.

DETAILED DESCRIPTION:
Efforts at treating radiation-induced cognitive and neuropsychiatric declines with medications have shown only minimal preliminary cognitive benefit and do not affect quality of life (QOL). Given the structural and functional brain alterations associated with WBRT, preventing rather than treating these radiation-induced changes may produce more favorable outcomes. Innovative radiotherapy techniques can limit the dose of radiation applied to specific brain structures without compromising tumor coverage. In this light, Radiation Therapy Oncology Group (RTOG) recently published a study evaluating the hippocampal avoidance whole brain radiation therapy (WBRT) in patients with brain metastases. They suggest potential preservation of cognitive function with this approach with no perceived detriment in survival. This concept is currently undergoing investigation in a definitive randomized controlled study (NRG-CC003) in patients receiving prophylactic cranial irradiation for small cell lung cancer. However, no other studies to date have prospectively evaluated avoidance of other particularly sensitive brain regions.

One brain region that has received little attention in the radiotherapy literature is the corpus callosum. The genu of the corpus callosum contains thin, densely packed neural fibers that primarily connect the prefrontal association areas and the anterior inferior parietal regions of the brain. Damage or thinning of the genu is associated with reduced functioning on tests of executive functioning, attention, working memory, processing speed, verbal fluency and memory in a variety of healthy and patient groups including aging, cerebral small vessel disease, traumatic brain injury, multiple sclerosis , human immunodeficiency virus, mild cognitive impairment secondary to Parkinson's disease, and euthymic bipolar disorder. The limited existing data in adults receiving WBRT for brain metastases suggest that they also perceive progressive declines in motivation following treatment. Given its apparent involvement in a wide range of cognitive processes, the genu of the corpus callosum is an excellent candidate for sparing in WBRT. This relatively small area has the potential to preserve cognitive functioning across several domains if guarded from the damaging effects of radiation. In this study patients will receive the standard whole brain radiation dose of 3000 centigray (cGy) in 10 fractions, but intensity modulated radiation therapy will be utilized to limit radiation dose to the genu of the corpus callosum. Patients will undergo cognitive testing at baseline and at 4-, 6- and 12-months following completion of brain radiation to evaluate the study hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof or unequivocal cytologic proof solid tumor malignancy. This may be obtained from either the primary or any metastatic site
* Mini Mental State Examination (MMSE) ≥24
* Age≥ 18 years
* Karnofsky Performance Status (KPS) ≥70
* Patient does not have metastases to the genu
* Patient must be scheduled to undergo treatment with whole brain radiation therapy (WBRT) to manage the brain metastases
* Patients of childbearing potential (male or female) must practice adequate contraception due to possible harmful effects of radiation therapy on an unborn child
* Patient must have the ability to understand and the willingness to sign a written informed consent document
* All patients must be informed of the investigational nature of this study and must be given written informed consent in accordance with institutional and federal guidelines
* Patient must have a minimal life expectancy of at least 6 months
* Patients receiving prior stereostatic radiosurgery (SRS) for brain metastases are eligible

Exclusion Criteria:

* Prior WBRT
* MMSE<24
* Patient has brain metastases in the genu
* Patients must not have a serious medical or psychiatric illness that would, in the opinion of the treating physician prevent informed consent or completion of protocol treatment, and/or follow-up visits.
* KPS<70
* Non-native English speakers will be excluded since patients often lose their faculty with the language they acquired second before their native language is affected in the context of cognitive decline. This could adversely affect performance on verbal cognitive tasks.
* Patients with absolute contraindication to MRI imaging are not eligible for the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2017-07-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Rate of change of cognitive function | 4 months
  Evaluate changes in cognition from baseline to 4 months following genu-sparing whole brain radiation therapy (GS-WBRT)

SECONDARY OUTCOMES:
Rate of change of white matter microstructure | 4, 6 and 12 months
  Evaluate change in white matter microstructure following GS-WBRT utilizing diffusion tensor imaging
Rate of change of cognition | 4, 6 and 12 months
  Evaluate changes in cognition from baseline to 4, 6 and 12 months following GS-WBRT
Time to brain metastasis | 4, 6 and 12 months
  Document development of brain metastases in the spared genu of the corpus callosum
Rate of change in QoL | 4, 6 and 12 months
  Document changes in QOL, neuropsychiatric symptoms, and functioning in patients receiving GS-WBRT from pre-treatment to 4, 6 and 12 months following GS-WBRT
Rate of change in other frontally-mediated functions | 4, 6 and 12 months
  Document the stability of other frontally-mediated cognitive functions in those receiving GS-WBRT from pre-treatment to 4, 6 and 12 months following GS-WBRT.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Redmond, MD, MPH, Principal Investigator — The SKCCC at Johns Hopkins
Locations (2):
- United States (2):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - The SKCCC at Johns Hopkins, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No